CLINICAL TRIAL: NCT02378584
Title: The Clinical Results After Frozen-thawed Healthy Blastocyst Transfer in Natural Cycle Versus Cycle With Endometrial Preparation
Brief Title: Natural Cycle Versus Endometrial Preparation for Healthy Blastocyst Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC1978MA
Record Dates: First submitted 2015-02-06; First posted 2015-03-04 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- natural cycle (Other): Ultrasound controls and endocrine blood test to asses the day of ovulation for embryo transfer
  Interventions: Other: embryo transfer
- hormonal cycle (Active Comparator): Ultrasound controls and endocrine blood test to asses the endometrium thickness for embryo transfer
  Interventions: Other: embryo transfer

INTERVENTIONS:
Other: embryo transfer — healthy blastocyst transfer in natural and hormonal cycle
  Other Names: drug adminstration, clinical controls

SUMMARY:
This study evaluates the difference in pregnancy rate transferring a healthy blastocyst in natural or artificial cycle.

DETAILED DESCRIPTION:
The aim of the study was to verify the implantation capacity and ongoing pregnancy rate of vitrified warmed euploid blastocyst in natural cycle versus endometrial artificial cycle with gonadotropin-releasing hormone (GnRH-agonist) pituitary suppression.

ELIGIBILITY:
Inclusion Criteria:

* frozen-thawed healthy blastocyst

Exclusion Criteria:

* post thawed not survival healthy blastocyst

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 236 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate confirmed by ultrasound evidence of fetal heart activity | 12 weeks after embryo transfer

SECONDARY OUTCOMES:
live-birth rate confirmed by the number of born | term pregnancy delivery
cost-benefit of two endometrial preparation protocol | 30 weeks beginning from day 21 of the previous cycle day up to the pregnancy test
  Assessment of drug cost and the count of clinical visit, laboratory dosages and venous sampling
The number of patients with the anxiety and depression increase | Six weeks beginning on the day of treatment start, on the day of progesterone administration, on the day of blastocyst transfer and the pregnancy test
  the psychological questionnaire (HADS) administered on four time point

CONTACTS AND LOCATIONS:
Overall Officials: ERmanno Greco, MD, Study Director — European Hospital
Locations (2):
- Italy (2):
  - European Hospital, Rome, RM
  - European Hospital, Rome, Roma

REFERENCES:
- [Derived] Greco E, Litwicka K, Arrivi C, Varricchio MT, Caragia A, Greco A, Minasi MG, Fiorentino F. The endometrial preparation for frozen-thawed euploid blastocyst transfer: a prospective randomized trial comparing clinical results from natural modified cycle and exogenous hormone stimulation with GnRH agonist. J Assist Reprod Genet. 2016 Jul;33(7):873-84. doi: 10.1007/s10815-016-0736-y. Epub 2016 May 24. PMID 27221477